CLINICAL TRIAL: NCT01009801
Title: A Phase I Open Label/Phase II Randomized, Double-Blind, Multicenter Trial Investigating the Combination of Everolimus and TransArterial ChemoEmbolization (TACE) With Doxorubicin in Patients With Hepatocellular Carcinoma
Brief Title: Transarterial Chemoembolization With Doxorubicin With or Without Everolimus in Treating Patients With Liver Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: due to slow patient recruitement.
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAKK 77/09; SWS-SAKK-77-09; SWS-SASL-30; EU-20986; CDR0000658353
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; recurrent adult primary liver cancer; localized resectable adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Doxorubicin; Everolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Active Comparator): Patients receive oral placebo once daily for up to 12 months and undergo TACE comprising doxorubicin-eluting beads as in phase I at the MTD.
  Interventions: Drug: doxorubicin-eluting beads; Other: placebo
- Arm II (Experimental): Patients receive oral everolimus once daily for up to 12 months and undergo TACE comprising doxorubicin-eluting beads as in phase I at the MTD.
  Interventions: Drug: doxorubicin-eluting beads; Drug: everolimus

INTERVENTIONS:
Drug: doxorubicin-eluting beads — Patients receive oral placebo or everolimus once daily for up to 12 months and undergo TACE comprising doxorubicin-eluting beads as in phase I at the MTD.
  Other Names: Adriamycin
Drug: everolimus — Patients receive oral everolimus once daily for up to 12 months and undergo TACE comprising doxorubicin-eluting beads as in phase I at the MTD.
  Other Names: RAD001
  Arms: Arm II
Other: placebo — Patients receive oral placebo once daily for up to 12 months and undergo TACE comprising doxorubicin-eluting beads as in phase I at the MTD.
  Arms: Arm I

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Chemoembolization kills tumor cells by carrying drugs directly into the tumor and blocking the blood flow to the tumor. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether transarterial chemoembolization with doxorubicin is more effective when given alone or when given together with everolimus in treating patients with liver cancer.

PURPOSE: This randomized phase I/II trial is studying the side effects and best dose of everolimus when given together with transarterial chemoembolization with doxorubicin and to see how well it works compared with giving transarterial chemoembolization with doxorubicin alone in treating patients with liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the recommended dose of everolimus in patients with hepatocellular carcinoma (HCC) treated with transarterial chemoembolization with doxorubicin-eluting beads (TACE). (Phase I)
* Determine the efficacy and tolerability of everolimus in patients with HCC treated with TACE as compared to TACE alone. (Phase II)

OUTLINE: This is a multicenter, dose-escalation phase I study followed by a randomized phase II study.

* Phase I: Patients receive oral everolimus once daily in the absence of disease progression or unacceptable toxicity. Beginning 7 days after the start of everolimus patients undergo transarterial chemoembolization (TACE) comprising doxorubicin-eluting beads into the hepatic artery followed in 4 weeks by an MRI. If viable tumor is found patients undergo another TACE treatment continuing every 4 weeks for up to 5 treatments.
* Phase II: Patients are stratified according to center, age (≤ 60 vs > 60 years), and number of lesions (≤ 3 vs > 3). Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive oral placebo once daily for up to 12 months and undergo TACE comprising doxorubicin-eluting beads as in phase I at the maximum tolerated dose (MTD).
  * Arm II: Patients receive oral everolimus once daily for up to 12 months and undergo TACE comprising doxorubicin-eluting beads as in phase I at the MTD.

In both arms, patients receive treatment for up to 12 months in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for analysis of AFP tumor markers. Patients also complete quality of life questionnaires, Health Economic Assessment, and EQ5D questionnaires at baseline and periodically during the study.

After completion of study treatment, patients are followed on day 30, and then every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically, cytologically, or radiologically confirmed hepatocellular carcinoma

  * Intermediate stage B (according to Barcelona Clinic Liver Cancer classification)
  * Child-Pugh score < 8
  * No tumor involvement > 50% of whole liver
* No advanced stage disease (i.e., either portal invasion [segmental portal obstruction] or extrahepatic spread)
* No presence or history of metastatic disease
* Candidate for transarterial chemoembolization after multidisciplinary discussion (tumor board)
* Not on an active waiting list for liver transplantation

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Hemoglobin ≥ 90 g/L
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Bilirubin ≤ 1.5 x upper limit of normal (ULN)
* ALT ≤ 4 x ULN
* INR ≤ 2
* Creatinine ≤ 1.5 x ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 12 months after completion of study therapy
* Negative pregnancy test
* None of the following contraindications:

  * Complete portal vein thrombosis
  * Large arterio-portal or arterio-venous fistula within the liver
  * Allergy to contrast media
  * Contraindication to hepatic artery catheterization, such as severe peripheral vascular disease precluding catheterization
* No active heart disease, including any of the following:

  * NYHA class II-IV congestive heart failure
  * Active coronary artery disease (myocardial infarction > 6 months prior to trial entry allowed)
  * Cardiac arrhythmias requiring anti-arrhythmic therapy (beta-blockers or digoxin permitted)
  * Uncontrolled hypertension
* No hypertension, defined as systolic blood pressure (BP) > 150 mm Hg or diastolic BP > 90 mm Hg despite optimal medical management
* No thrombotic or embolic events within the past 6 months including any of the following:

  * Cerebrovascular accident (including transient ischemic attacks)
  * Pulmonary embolism
  * Deep vein thrombosis
* No serious non-healing wounds, including wounds healing by secondary intention, acute or non-healing ulcers, or bone fractures within 3 months of fracture
* No evidence of bleeding diathesis
* No history of hemoptysis
* No clinically serious infection > grade 2 (NCI CTCAE Version 3.0) except for HBV and HCV infection
* No known HIV infection
* No CTCAE acute adverse events grade > 2 after prior TACE therapy
* No other prior or concurrent malignancy that is distinct in primary site or histology from HCC, except carcinoma in situ of the cervix, treated nonmelanoma skin cancer, superficial bladder tumor (Ta, Tis, T1), or any cancer curatively treated > 3 years prior to entry
* No psychiatric disorder precluding understanding of information on trial related topics, giving informed consent, filling out QL forms, or interfering with compliance for oral drug intake
* No serious underlying medical condition, at the judgment of the investigator, which could impair the ability of the patient to participate in the trial (e.g., active autoimmune disease, uncontrolled diabetes)
* No known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs
* No contraindication to have MRI (e.g., pacemaker)
* No organ allograft
* No known impairment of swallowing that would preclude administration of everolimus
* Completed baseline quality of life, BL-HEA, and EQ5D questionnaires (Phase II only)
* Able to comply and have geographic proximity to allow proper staging and follow-up

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior transarterial embolization/chemoembolization [limited to 5 treatments], radiofrequency ablation, cryoablation, radiation therapy or percutaneous ethanol injection
* At least 4 weeks since prior sorafenib
* At least 30 days since treatment with other experimental drugs or other anticancer therapy, or treatment in another clinical trial
* At least 30 days since use of biologic response modifiers (e.g., G-CSF and other hematopoietic growth factors)
* More than 4 weeks since prior and no concurrent major surgery
* More than 3 weeks since prior and no concurrent radiotherapy
* Concurrent erythropoietin allowed provided no dose adjustment is undertaken within 1 month prior to the trial or during the trial
* No concurrent anticancer drugs (e.g., bevacizumab, and any drugs that target VEGF or VEGF receptors)
* No concurrent investigational drugs
* No concurrent known strong CYP3A4 inhibitors (e.g., ketoconazole, fluconazole, itraconazole, voriconazole, erythromycin, clarithromycin, diltiazem, verapamil, and protease inhibitors)
* No concurrent known strong CYP3A4 inducers (e.g., carbamazepine, continuous treatment with dexamethasone [> 2 mg/day for > 7 days], phenobarbital, phenytoin, rifampicin, and St. John's wort)
* No concurrent grapefruit, grapefruit juice, and products containing bitter oranges
* No concurrent systemic corticosteroids (e.g., > 1 mg/kg prednisolone) for more than 2 weeks
* No concurrent angiotensin converting enzyme inhibitors (ACE-I)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (Phase I) | after 6 weeks from registration
  Dose limiting toxicity (DLT) (observed within the first TACE period)
Time to progression (Phase II) | 12 weeks after randomisation

SECONDARY OUTCOMES:
Time to progression (Phase I) | 12 weeks after registration
Progression-free survival (Phase II) | Time from randomization until event occurs (see description):
  * Relapse or progression assessed according to the modified RECIST criteria
  * Death of any cause
  * Metastasis outside of liver
Progression-free survival at 12 months (Phase II) | within 12 months after randomisation
Tumor response according to adapted RECIST criteria (Phase II) | during treatment
Overall survival (Phase II) | Time from randomisation until death from any cause
Response duration (Phase II) | See description
  From the time when criteria for response (CR or PR) are met, until documentation of relapse or progression thereafter.
Time to treatment failure (Phase II) | See description
  Time from registration to any treatment failure including disease progression or premature (within 12 months) discontinuation of treatment for any reason (e.g., disease progression, toxicity, patient preference, initiation of new treatment without documented progression, Initiation of second line of TACE, Initiation of sorafenib therapy or death).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Dufour, MD, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (8):
- Switzerland (8):
  - Inselspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Clinica Luganese di Moncucco, Lugano
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Institut Central des Hopitaux Valaisans / Hôpital de Sion, Sion
  - UniversitaetsSpital Zuerich, Zurich